CLINICAL TRIAL: NCT03672201
Title: Standardizing Care for Neuropsychiatric Symptoms and Quality of Life in Dementia
Acronym: StaN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University of Calgary (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); Douglas Mental Health University Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1482
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer's Disease; Alzheimer Dementia (AD); Aggression
Keywords: Aggression; Agitation; Alzheimer's disease; Integrated Care Pathway; StaN; Dementia
MeSH Terms: conditions — Alzheimer Disease; Aggression; Psychomotor Agitation; Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and assessors will be blind to the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Integrated Care Pathway (ICP) Arm (Active Comparator): The ICP consists of 1) a cleanup phase during which a thorough assessment of pharmacotherapy to discontinue unnecessary medications, is performed; 2) Structured non-pharmacological interventions, which would have started as soon as randomization occurred and would continue before any pharmacological intervention for 2 weeks as stand-alone interventions; and 3) a pharmacological intervention phase: in this phase the medications algorithm for AD-AA is initiated.
  Interventions: Behavioral: Non-Pharmacological Intervention; Other: Pharmacological Intervention
- Treatment-As-Usual (TAU) Arm (No Intervention): Following eligibility and baseline assessments, half of the participants will be randomized to TAU. TAU will consist of the typical care that the interdisciplinary team provides at each site for AD-AA. No predetermined cleanup phase, non-pharmacological interventions, algorithmic pharmacological interventions will be systematically part of TAU.

INTERVENTIONS:
Behavioral: Non-Pharmacological Intervention — The behavioural intervention will be a structured implementation of individualized activities to be followed and customized as per the needs of the participant.
  Other Names: Behavioural Intervention
  Arms: The Integrated Care Pathway (ICP) Arm
Other: Pharmacological Intervention — The medication algorithm provides recommendations to the treatment team about algorithmic treatment and assessments as per the ICP but ultimately the decision to prescribe any particular intervention will be the treatment team's decision and the recommendations of the research team for ICP arm will not be binding for the treatment team.
  Arms: The Integrated Care Pathway (ICP) Arm

SUMMARY:
The object of this study to evaluation an Integrated Care Pathway (ICP) to treat Aggression and Agitation in Alzheimer's disease (AD-AA). The ICP is an algorithmic approach to use psychotropic medications and non-pharmacological interventions based on standardized assessments which fosters measurement-based decision making. This study will assess the efficacy of the ICP to treat AD-AA and its impact on inappropriate use of medications in inpatient settings and Long-Term Care Facilities (LTCF).

The investigators will enroll and randomize 220 participants with AD-AA (110 inpatient and 110 LTCFs) to ICP vs. Treatment As Usual. Further, this study will also examine the impact of the ICP on caregiver burden and undertake a cost-effectiveness analysis of the ICP for patients with AD-AA.

DETAILED DESCRIPTION:
This project will take place in 7 sites across two settings: Inpatient (CAMH in Toronto, Douglas Hospital Research Centre in Montreal, Parkwood Institute in London, and the University of Calgary in Calgary); and LTCFs affiliated with CAMH in Toronto and Parkwood Institute in London.

After a project initiation phase of 6 months, the investigators will enroll and randomize 220 participants with AD-AA (110 inpatient and 110 in LTCFs) to ICP vs.TAU. In this randomized control trial (RCT) phase of the project, participants will be treated for 12 weeks. There will be two primary outcome measures: (i) the Cohen-Mansfield Agitation Inventory (CMAI) Total Frequency Score (CMAI-frequency) and (ii) the proportion of participants on polypharmacy. These measures will be conducted at baseline, end of non-pharmacological intervention phase, the mid-point of pharmacological interventions and end of RCT. Neuropsychiatric Inventory-Questionnaire (NPI-C) will be used to assess global burden of neuropsychiatric symptoms at baseline, end of non-pharmacological intervention phase and exit. The modified Clinical Global Impression of Change (CGIC) will also be measured at predetermined time points throughout the 12 weeks to determine response as defined by CGIC < 3. CGIC is a 7-point Likert scale to rate each patient along a continuum from marked improvement to marked worsening, based on global clinical impression. Rating of < 3 indicates moderate or marked improvement in agitation as compared to baseline. At the end of the RCT, each participant will be naturalistically followed up for an additional 6 months during which the investigators will collect both clinical and health economics data from the Institute for Clinical Evaluative Sciences (ICES) database. The RCT phase will be completed after 18 months, and during the last part of this project, the investigators will analyze the data from the RCT and complete all naturalistic follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of Dementia of Alzheimer's or Mixed type using the Diagnostic and Statistical Manual of Mental Disorders, 5th Ed. (DSM-5) criteria
2. AD-AA as defined by Agitation in cognitive disorders; International Psychogeriatric Association provisional consensus clinical and research definition
3. Participant or substitute decision maker (SDM) able and willing to provide consent for enrollment in the study
4. 50 years or older
5. Medical stability to participate in the trial.

Exclusion Criteria:

1. Having dementia other than Alzheimer's or Mixed type.
2. DSM-5 diagnoses other than dementia that is thought to be significantly impacting the presentation of AD-AA such as delirium, bipolar disorder, or major depressive disorder.
3. Any other reason which in the opinion of study investigator will make the study participation intolerable for the participant.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cohen-Mansfield Agitation Inventory - Total Frequency Score (CMAI - Frequency) | Conducted at baseline, 3 weeks, 8 weeks, and 12 weeks
  The Cohen-Mansfield Agitation Inventory (CMAI) Frequency score measures burden of agitation in patients with dementia. CMAI-frequency score ranges between 29 to 203, higher scores indicate worsening of symptoms.
The proportion of participants on polypharmacy | Data collected at baseline, 3 weeks, 8 weeks, and 12 weeks
  The percentage and the total number of participants on 2 or more psychotropics

SECONDARY OUTCOMES:
The impact of the ICP on falls | Every 2 weeks
  Recording the number of falls

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Rajji, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (6):
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - Providence Care, Kingston, Ontario
  - LAWSON Health Research Institute, London, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario
  - Ontario Shores Centre for Mental Health Sciences, Whitby, Ontario
  - Douglas Hospital Research Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choudhury S, Colman S, Chu L, Davies SJC, Derkach P, Elmi S, Fischer CE, Gerretsen P, Graff-Guerrero A, Hussain M, Ismail Z, Khan SS, Kim D, Krisman L, Moghabghab R, Mulsant BH, Nair V, Pollock BG, Rej S, Rostas A, Streiner D, Van Bussel L, Rajji TK, Kumar S, Burhan AM; StaN Study Group. Sex Differences in Phenomenology of Behavioral and Psychological Symptoms of Dementia. Neurodegener Dis. 2025 Oct 2:1-11. doi: 10.1159/000548713. Online ahead of print. PMID 41037500
- [Derived] Tavakoli E, Niciforos E, Amid P, Cuperfain AB, Burhan AM, Colman S, Chu L, Davies SJC, Derkach P, Gerretsen P, Graff-Guerrero A, Hussain M, Ismail Z, Kim D, Krisman L, Mulsant BH, Pollock BG, Rej S, Rostas A, Rajji TK, Van Bussel L, Kumar S, Elmi S. The impact of lifetime excessive alcohol use on behavioural and psychological symptoms of dementia. Alcohol Alcohol. 2025 Jul 16;60(5):agaf048. doi: 10.1093/alcalc/agaf048. PMID 40794901
- [Derived] Zarei S, Colman S, Rostas A, Burhan AM, Chu L, Davies SJ, Derkach P, Elmi S, Hussain M, Gerretsen P, Graff-Guerrero A, Ismail Z, Kim D, Krisman L, Moghabghab R, Mulsant BH, Nair V, Pollock BG, Rej S, Simmons J, Van Bussel L, Rajji TK, Kumar S; StaN Study Group. The Rationale and Design of Behavioral Interventions for Management of Agitation in Dementia in a Multi-Site Clinical Trial. J Alzheimers Dis. 2022;86(2):827-840. doi: 10.3233/JAD-215261. PMID 35147535